CLINICAL TRIAL: NCT01027130
Title: Haptoglobin and Preeclampsia
Status: Completed | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Other Study IDs: HAPPET
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy control: 240 female subjects without preeclampsia
- preeclampsia: 120 female subjects with preeclampsia

SUMMARY:
The purpose of this study is to show that a certain protein called haptoglobin protects against preeclampsia which is a common pregnancy complication.

ELIGIBILITY:
Inclusion Criteria:

* all women

Exclusion Criteria:

* women with hypertension

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: women coming to give birth at our medical center
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai-Zion Medical Center, Haifa, Israel